CLINICAL TRIAL: NCT04031300
Title: Performance and Safety Evaluation of a Novel Non-invasive Glucose Monitoring Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to change in project strategy (new intended use)
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RSP-20
Record Dates: First submitted 2019-03-26; First posted 2019-07-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSP-20 (Experimental): Subjects will perform daily measurements on the IMD (Prototype 0.5) in addition to capillary reference measurements for 48 days.
  Interventions: Device: Prototype 0.5

INTERVENTIONS:
Device: Prototype 0.5 — Investigational Medical Device collecting spectral Raman data non-invasively from tissue
  Other Names: P0.5

SUMMARY:
This pivotal multicenter study has been launched to collect spectral Raman data paired with validated glucose reference values in diabetic patients.

DETAILED DESCRIPTION:
Participants will be enrolled at six different sites in four different countries. All participants will undergo identical procedures, which include four steps: Baseline visit (1 day), calibration period (25 days), validation period (23 days) and a close-out visit (1 day) with a total duration of 50 days.

The calibration period consists of 23 home-based days and two in-clinic days. At the two in-clinic days, measurement sessions are performed every 30 minutes. A measurement session consists of two reference measurements (Contour Next One) and three measurements on the Investigational Medical Device. The glucose level of the participants is manipulated by administration of a glucose rich drink. At home-based days, the subject must perform four measurement sessions a day. During the validation period, participants perform up to four home-based measurement sessions a day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Diagnosed with diabetes, all types except gestational diabetes
* Skin phototype 1-4
* Willing to perform a minimum of 8 finger sticks during each day of home-based measurements and 30 finger sticks at the two in-clinic study days
* Subject has a wireless internet connection at home to be used in the study

Exclusion Criteria:

* For female subjects: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* For female subjects: Breastfeeding
* Subject currently participating in another study
* Subject not able to understand and read the local language
* In investigator's opinion, subject is not able to follow instructions provided and as specified in the protocol
* Subject not able to hold hand/arm steady (including tremors and Parkinson's Disease)
* Subject diagnosed with cardiovascular diseases
* Reduced circulation in right hand evaluated by Allen's test
* Subjects receiving anticoagulants, active cancer treatment, tetracyclines and other medication/topical agents increasing photosensitivity
* Radiotherapy for the past six months
* Extensive skin changes, tattoos or diseases on right hand thenar (probe application site)
* Known allergy to medical grade alcohol used to clean the skin
* Medical history or any condition that may, in the opinion of the investigator compromise the subject's ability to participate
* Comorbidity or concomitant medical condition which, in the opinion of the Investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement accuracy | 6 months
  Accuracy of measurements performed on the IMD will be evaluated by data from subjects. Data will be analyzed by Mean Absolute Relative Difference (MARD).
Safety evaluation: paucity of adverse events | 6 months
  Safety of the IMD will be evaluated in a descriptive manner by the paucity of adverse events reported during the clinical study

SECONDARY OUTCOMES:
Device deficiencies | Up to 6 months
  Description of device deficiencies will be listed. Deficiencies will be reported during the clinical study.
Device usability | 6 months
  The use of the device will be evaluated by means of questionnaires. The subjects are asked if they encountered any problems during measurements, and if so, to elaborate the problems encountered.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (6):
- Denmark (2):
  - Steno Diabetes Center Copenhagen (SDCC), Gentofte Municipality
  - Steno Diabetes Center Odense (SDCO), Odense C
- Institut für Diabetes-Technologie Forschungs- und Entwicklungs-gesellschaft mbH an der Universität Ulm (IDT), Ulm, Germany
- Sweden (2):
  - Sahlgrenske University Hospital (SUH), Gothenburg
  - Department of Medicine, Uddevalla Hospital (UVH), Uddevalla
- University Hospitals Birmingham (UHB), Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No